CLINICAL TRIAL: NCT02032355
Title: The Feasibility of PetCO2 Prediction Hypotension Under Spinal Anesthesia for Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Geng guiqi (Other)
Responsible Party: Sponsor-Investigator, Geng guiqi, professor, Fudan University
Organization: Fudan University (Other)
Other Study IDs: 61538
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Hypotension; Carbon Dioxide
MeSH Terms: conditions — Hypotension | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- hypotension
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia

SUMMARY:
Maternal hypotension is a common side effect after spinal anesthesia for cesarean delivery.Decreased vascular resistance and cardiac output, due to sympathetic blockade1and blood pooling in blocked areas of the body respectively, are main causes of spinal anaesthesia-induced hypotension during Caesarean delivery.

Cardiac output, which has shown to be a better predictor of organ and placental perfusion than arterial blood pressure.Few studies have measured CO after spinal anesthesia in the maternal population.This is largely because of the lack of availability of accurate and reproducible noninvasive measurement techniques. Up to now, preventing hypotension has continued to focus on arterial blood pressure variables, fluid, and ephedrine requirements as markers of cardiovascular status, because these are more easily measured.

Investgators hypothesized that CO and PetCO2, in parturients with the degree of hypotension during spinal anaesthesia, would also have a positive and significant association.

ELIGIBILITY:
Inclusion Criteria:

* full-term gestation (>36 and <41 weeks of gestation) with a singleton pregnancy

Exclusion Criteria:

* emergency cases
* placenta praevia
* preeclampsia
* cardiovascular or cerebrovascular disease
* morbid obesity with a BMI≥40
* contraindications to spinal anaesthesia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: American Society of Anesthesiologists physical status I and II patients undergoing elective cesarean delivery under combined spinal-epidural (CSE) anesthesia
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
value of PetCO2 and changes in artery pressure | up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics & Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China